CLINICAL TRIAL: NCT04976998
Title: Role of Ultrasonography in the Diagnosis of Carpal Tunnel Syndrome and Detection of Its Severity
Brief Title: Role of Ultrasonography in the Diagnosis of Carpal Tunnel Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Ahmed Mohamed, radiological resident, Sohag University
Other Study IDs: Soh-Med-21-07-17
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Diagnostic Imaging; Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: those with symptoms of CTS
  Interventions: Diagnostic Test: imaging
- control group: normal people those with no symptoms of CTS
  Interventions: Diagnostic Test: imaging

INTERVENTIONS:
Diagnostic Test: imaging — imaging by ultrasonography and nerve conduction studies will be done for both grups
  Other Names: nerve conduction studies

SUMMARY:
This prospective study aims to evaluate the median nerve in Carpal Tunnel Syndrome by high-frequency ultrasound and color Doppler in comparison with clinical and Nerve conduction studies.

DETAILED DESCRIPTION:
This prospective study aims to evaluate the median nerve anatomical changes in Carpal Tunnel Syndrome by high-frequency ultrasound and color Doppler in comparison with clinical and Nerve conduction studies physiological changes to determine the efficacy of ultrasound to diagnose and determine the severity of carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Any Age Group with symptoms, clinical signs and NCS consistent with CTS

Exclusion Criteria:

* Uncooperative Patients .
* Patients with History of previous wrist surgery, fracture or traumatic nerve injury

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: sohag university hospital patients and attendants
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-08-29 (Estimated); Primary Completion 2022-02-02 (Estimated); Study Completion 2022-03-20 (Estimated)

PRIMARY OUTCOMES:
anatomical changes in the median nerve in carpal tunnel syndrome | imaging within 24 hours from the nerve conduction studies and clinical assessment of the patient
  compare the anatomical changes observed by ultrasonography in patients diagnosed with carpal tunnel syndrome and comparing the results with clinical and nerve conduction studies results

CONTACTS AND LOCATIONS:
Overall Officials: mostafa mm mohamed, MBBCH, Principal Investigator — Sohag University
Locations (1):
- Sohag University - Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided